CLINICAL TRIAL: NCT02585063
Title: Independent Prescribing Optometrists in Acute Ophthalmic Services
Status: Completed | Type: Observational
Sponsor: Aston University (Other)
Collaborators: Manchester Royal Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DT001
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Eye Abnormalities
Keywords: independent prescribing,; optometrist; acute care
MeSH Terms: conditions — Eye Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dual assessment: Where there is time and space, participants will be allocated to have a clinical assessment by the IP optometrist during their wait for the clinical assessment with the ophthalmologist. Both clinical assessments are needed to obtain measurement of agreement. There is no intervention. but participants have two clinical assessments rather than just one.

SUMMARY:
The UK government's Crown report titled 'Review of prescribing, supply & administration of medicines' enabled optometrists to train for the qualification of independent prescribing (IP). The UK introduced IP for optometrists in 2009. The proposed research focuses on the role of IP optometrist in the acute ophthalmic services of Manchester Royal Eye Hospital (MREH). The study will compare IP optometrists to consultant ophthalmologists in the ability to diagnose, manage and prescribe medication for patients accessing these services.

To achieve this comparison consenting participants will first have a clinical assessment with the IP Optometrist, where findings including diagnosis and management plan will be recorded onto a research proforma. The consultant ophthalmologist will be masked to the IP Optometrist's research proforma to prevent bias. The consultant ophthalmologist will then perform a clinical assessment on a second proforma and inform the participant of their diagnosis and management plan. Percentage agreement, kappa (κ) and weighted κ will be calculated for a range of parameters between the two proformas. Disagreement in diagnosis or management will be arbitrated by a separate ophthalmologist participating in the study with a specialty relevant to the participant's condition.

The main objective of the research is to expand the limited base of evidence of of IP optometrists' ability to diagnose, manage and prescribe medication and to determine whether they work at least as safely and effectively as consultant ophthalmologists in acute ophthalmic services. It is the first study in this area since the advent of IP for optometrists, with only one previous study published before IP was introduced. The research will enable the type and frequency of conditions presenting in these services to be measured. Furthermore it will identify conditions that IP optometrists can manage independently and enable guidelines for these conditions to be developed.

DETAILED DESCRIPTION:
What are the purpose and objectives of the research?

The primary aim of this prospective, masked, controlled comparative study is to measure the agreement in diagnosis between IP optometrists and the reference standard of consultant ophthalmologists.

A secondary aim is to measure agreement in management of the diagnosis, including the decision whether or not to prescribe medication. The choice of not prescribing medication is an important prescribing decision and will be counted as such. This measure is the novel aspect of the research as it provides evidence of IP optometrists' ability to safely prescribe.

What is the scientific justification for the research?

The NHS's emergency services are experiencing increasing demand (Ismail et al 2013), which is also true of MREH's Acute Referral Centre where IP optometrists work as part of a multidisciplinary team. There is a scientific need to provide an evidence base to validate and support the role of optometrists working in acute ophthalmic services, as well as provide evidence of IP optometrist's ability to safely prescribe medication. This evidence base may in turn lend support to nationally extending the role of IP Optometrists' and their skills to the benefit of the Health Service. Establishing an audit meets the clinic need to monitor performance of IP optometrists working in this extended role. Guidelines for IP optometrists working within MREH Acute Ophthalmic Services offer a way to optimise the running of the clinic as patient can be triaged to clinicians and ophthalmologists feed to see complex cases.

A novel aspect of this study is that it will compare optometrists' management decisions involving the prescribing of ocular medication since IP was introduced (General Optical Council 2014). There is no evidence of studies into the safety of such prescribing decisions by IP optometrists in acute ophthalmic care. Hau et al (2007) study entitled 'An evaluation of optometrists' ability to correctly identify and manage patient s with ocular disease in the accident and emergency department of an eye hospital' was before the introduction of IP.

Duration

The study will begin in Summer 2015, pending ethics approval, and will last for 18 months.

Sample size

A sample of up to 1500 may be achieved based on 20 participants per week over a period of 18 months. This breaks down to 2.5 participants per study session. It is anticipated that the principal IP optometrist of the Acute Referral clinic who works there 4 sessions a week will have the potential to perform ~690 clinical assessments for the study. The remaining three IP optometrists who work one session a week will have the potential to perform ~172 clinical assessments.

A sample size of 500 with disagreement on diagnosis in 15 individuals is required to give a target disagreement rate of 3.0% (binomial 95% CI 1.7-4.9%). The larger anticipated sample size will ensure that at least 500 are available where a prescribing decision has been made, whilst maintaining small binomial confidence intervals.

Method

The protocol for the study is as follows:

1. Recruitment Patients will be invited to take part in the study and given the study information either while being triaged in the walk-in, nurse-led Emergency Eye Centre (EEC) to the appointments-based Acute Referral Clinic (ARC) or at arrival at ARC. An approved poster will advertise the study and will be place on the wall in both ARC and EEC. There will be a smaller version on the reception desk at both ARC and EEC accompanied by a participant information leaflet.

   Willingness to participate may depend on the individual and their presenting complaint. It may be expected that someone with severe symptoms who is triaged to be seen more urgently would be less inclined to have two clinical assessments. Analysis of the presenting complaints may identify trends in the severity versus participation in the study. It will be made clear that there is no obligation to participate and that if people do decide to take part that they can withdraw at any time.
2. Informed consent There are aspects about the way that the data will be used that warrants the consent of participants, with adequate assurance that privacy and confidentiality will be maintained. All participating optometrists and ophthalmologists will take informed consent. The clinicians will be trained in Good Clinical Practice and taking informed consent. Consent may take place during the 4 hour wait in the clinic or upon returning for a follow up appointment where appropriate (participants can only have the comparative clinical assessments once to ensure masking).
3. Participant allocation and capping Where there is time and space, participants will be allocated to have a clinical assessment by the IP optometrist during their wait for the clinical assessment with the ophthalmologist. Both clinical assessments are needed to obtain measurement of agreement.

   Sessions where a Consultant Ophthalmologist is in ARC will be allocated as a 'study session'. The study sessions will need to be allocated to ensure that approximately equal numbers of patients will be seen by the participating IP Optometrists. Consultant ophthalmologists with various specialties work with IP optometrists across 8 half day clinics during the week. A limitation of collecting data from these set times is that if there are conditions specific to presenting on an evening or weekend they will not be sampled representatively. Whilst this restricts analysis of certain conditions it ensures the focus of the study, evaluation of management by IP Optometrists to be achieved.

   A pragmatic approach will be required for the recruitment of patients into the study given organisational issues or limited time and rooms available to see patients. The recruitment per session for the comparative arm of the study can be capped by the Ophthalmologist within the clinic. Allowing a cap ensures that waiting times are kept within reason and the level of care is maintained. The cap risks introducing selection bias as potential participants presenting to clinic early may be more likely to be have the two comparative clinical assessments. The time of attendance in clinic will be recorded to monitor if this happens.
4. IP optometrist's clinical assessment The following protocol is relevant for participants undergoing the two comparative clinical assessments. The IP optometrists will receive the patient's notes, temporary if presenting on the day, or full notes if attending a follow up. There may be nursing notes including from the same day including the following; patient history record of measured vision or visual acuity (including pin hole visual acuity where it is reduced to 0.20logMAR or less), findings from an assessment by slit-lamp of the front of the eye, measurement of intraocular pressure, a record of pupil reaction and time of pupil dilation where appropriate.

   The consultation will be documented on the study proforma and include the following:
   * history and symptoms including where appropriate; medical history, medication, previous ocular history, family history, occupation, driving status.
   * examination of the anterior segment of the eye by slit-lamp or direct ophthalmoscopy.
   * examination of the posterior segment where appropriate by direct ophthalmoscopy or indirect biomicroscopy
   * tonometry (if not previously recorded)
   * other diagnostic tests as needed (e.g. pachymetry, colour vision).

   The assessment is expected to lead to the formation of a working diagnosis and management plan including the following where appropriate; prescribing ophthalmic medication, follow-up, referral or discharge. The proforma will have boxes to record diagnosis (primary and secondary where appropriate), management plan, treatment (including strength and dosing regimen), advice to patient and in addition a comments box to permit a judgment on whether the case could have been managed solely by an IP Optometrist. There may be occasions where conditions present outside of the scope of the IP Optometrists experience, which will be recorded in the comments box noting any reasons for this.
5. Masking and storage IP optometrist's proforma The first study proforma will be filed into one drawer of a cabinet in a lockable office. The proformas will be returned to the patient notes after the ophthalmologists assessment has concluded and anonymous photocopies taken of both proformas by the research optometrist (or where there is absence or holidays a different IP optometrist to ensure masking).
6. Ophthalmologist's clinical assessment The ophthalmologist will receive their own copy a proforma along with the patient's notes, but remain masked to the IP optometrist's assessment. They will follow the same protocol and then confirmation of participant's diagnosis and management plan.
7. Masking and storage of ophthalmologists proforma The ophthalmologist's proforma will be securely stored in a separate drawer in the lockable office. The proforma will be returned to the patient notes after anonymous copies of the proforma are photocopied by the end of the clinical session.
8. Storage of data Daniel Todd will analyse the anonymous copied proformas and keep the data stored securely to adhere to the legal requirement of data protection. Proformas will be kept in secured locked office and electronic data will be encrypted and stored on secure NHS computer.
9. Statistical analysis of agreement The results of the IP Optometrists' proformas compared for agreement in diagnosis (primary outcome) and management including prescribed medication (secondary) against the consultants' proforma. Percentage agreement, kappa (κ) and weighted κ will be calculated for a range of parameters. A system adapted by Marks et al (2012) in a comparative of study between ophthalmologists and optometrist in glaucoma management, which is originally based one by Banes et al (2006) will be employed where the following scores are given; 1.00 = agreement, 0.75 = 1 step from agreement, 0.50 = 2 steps from agreement, 0.25 = 3 steps from agreement and 0.00 = 4 steps of more. Agreement between diagnoses and clinical management plans would support IP Optometrist's role in the field and provide evidence of their ability to safely prescribe.
10. Arbitration of disagreement An arbitrator will confirm where there is disagreement; it may be that several diagnoses apply or different ways of prescribing are acceptable. Arbitration refers to assessment of agreement and not to the clinical care provided. Disagreement will be confirmed by showing a participant's notes and proformas to the arbitrator, who is a second ophthalmologist participating in the study specialty relevant to the participant's complaint. The arbitrator would provide their diagnosis and management plan while being masked to those reached by the IP optometrist and first ophthalmologist. Weekly meeting with each arbitrator will be arranged by Daniel Todd.
11. Dissemination of results Once the study's data has been collected and analysed then discussion and conclusions will be published. Where participants have expressly requested feedback from the study, they will be informed as requested (by telephone, e-mail or letter).

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients referred to MREH's Acute Referral Clinic. Referrals to ARC may be by MREH's nurse led Emergency Eye Centre, by optometrists in the community, by general practitioners, by other medical specialist or by patients with known uveitis (an inflammatory eye condition that may be recurrent).
2. Adult patients invited within the Emergency Eye Centre.
3. Adult patients with capacity for informed consent and willingness to participate.
4. Adult patients who are English speaking.

Exclusion Criteria:

1. Patients under the age of 18 years.
2. Patients without capacity or willingness to consent.
3. Patients unable to comply with routine clinical ophthalmic assessments.
4. Patients who require an interpreter.
5. Patients presenting with conditions that require immediate intervention for example; chemical burn or acute angle closure glaucoma.
6. Patients who are prisoners or young offenders.
7. All in-patients as their care is outside of the skills and experience of an optometrist.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be invited to take part in the study and given the study information either while being triaged in the walk-in, nurse-led Emergency Eye Centre (EEC) to the appointments-based Acute Referral Clinic (ARC) or at arrival at ARC. An approved poster will advertise the study and will be place on the wall in both ARC and EEC. There will be a smaller version on the reception desk at both ARC and EEC accompanied by a participant information leaflet.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Prescribing decision | Through study completion - up to 18 months
  The prescribing decisions of ophthalmologists and optometrists will be compared. They will be documented via self-reports.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tromans, PhD, Study Chair — Manchester Royal Eye Hospital
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom